CLINICAL TRIAL: NCT01491646
Title: Integrated Diagnostics Characterization of Right Ventricular Diastolic Flow Dynamics in Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Siemens Medical Solutions (Industry)
Responsible Party: Sponsor
Other Study IDs: HS 2512
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; cardiac magnetic resonance imaging; Characterize and quantify RV vortex flow; Assess feasibility of cardiac MR for RVDD diagnosis; Biomarker information to help diagnose
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — plasma, serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Pulmonary Hypertension: Previous diagnosis of PH by right heart catheterization
- Healthy Controls: Healthy controls without lung/heart conditions

SUMMARY:
Pulmonary hypertension (PH) is a condition in which high blood pressure develops in the lungs and right side of the heart. People with PH suffer from shortness of breath, chest pain, heart failure, heart rhythm problems, and fainting. PH is diagnosed using a test called a cardiac catheterization where blood pressure is measured directly using a tube placed in the right side of the heart and lung arteries. Because a cardiac catheterization is invasive, researchers are investigating ways to diagnose PH using imaging tests that are not invasive. The study will evaluate whether or not a magnetic resonance image (MRI) of the heart, and blood tests can detect PH.

DETAILED DESCRIPTION:
The adaptive changes that result from chronic pressure overload in pulmonary arterial hypertension (PAH) lead to myocardial hypertrophy, stiffening, and right ventricular diastolic dysfunction (RVDD). A growing body of evidence has identified RVDD as an important prognostic indicator for PAH.1 Diagnosis of RVDD relies upon 1) elevated brain natriuretic peptide (BNP), which correctly identifies RVDD in the PAH population but remains a nonspecific marker, and 2) echocardiography, as defined by reduced early (E') tricuspid annular velocity, elevated ratio of early filling tricuspid inflow peak velocity to E' (E/E'), and prolonged relaxation time (RT). 2 However, the right ventricle's unusual anatomy and susceptibility to altered loading conditions have raised questions about the ability of echo indices to accurately reflect complex diastolic mechanics. The development of a robust non-invasive application for RV diastolic assessment may improve the understanding, diagnosis, and management of RVDD and therefore PAH.

Similar to the left ventricle, rheological analysis of right ventricular inflow in canine models has identified the formation of diastolic vortex rings.3 Vortex rings develop from high velocity diastolic jet emanating from the valvular annulus interacting with stationary blood in the ventricle. Vortex ring formation time has successfully identified left ventricular diastolic dysfunction.4 Numerous additional vortex properties exist, including depth, transverse position, length, width, and sphericity index, that offer novel and robust diastolic flow characterization with the potential incremental diagnostic value to existing echo parameters. Vortex formation and analysis in RVDD has yet to be studied.

Vortex measurement can be performed using dimensional (4D) (time-resolved three-dimensional) cardiac MRI (CMR). 4D CMR captures the complex multidirectional nature of flow through volumetric rendering of fluid vectors and velocity using blood flow streamlines and particle traces. In contrast to echocardiography, 4D CMR is not limited by poor acoustic windows commonly seen in patients with respiratory disease and PAH, making it an ideal noninvasive modality for vortex characterization.

The biological adaptations resulting from chronic pressure overload in PAH might be correlated to the blood levels of different categories of biomarkers. They might play a role in the screening, diagnosis, monitoring or prognosis of patients with PAH and RVDD. Special mention can be made to the natriuretic peptides (BNP, NT-proBNP) based on their clinical value as hemodynamic markers in congestive heart failure. Cardiac markers of necrosis (asTroponin-I, and particularly the high sensitivity assays) might identify even minimal areas with such myocardial cell damage. The biological evaluation of cardiac fibrosis, might be assessed by markers of fibrosis, as Hyaluronic acid (HA), Procollagen III amino terminal peptide (PIIINP) and Tissue inhibitor of metalloproteinase 1 (TIMP-1). The potential role of the inflammatory component, can be evaluated with MPO (myeloperoxidase, pro-inflammatory enzyme), IL-6 (pro-inflammatory cytokine), C-RP (C-reactive protein)

The present study aims to:

1. Characterize and quantify RV vortex flow in normal subjects and PAH subjects with RVDD
2. Assess the feasibility of 4D CMR right ventricular diastolic vortex analysis for diagnosis of RVDD Hypothesis: 4D CMR vortex analysis accurately identifies RVDD, and the information provided by biomarkers helps by adding diagnostic information.

ELIGIBILITY:
Inclusion Criteria:

* previous diagnosis of PH by right heart catheterization
* RV diastolic dysfunction by echo
* normal RV systolic function
* age 18-75 years old
* no contraindication to MRI

Exclusion Criteria:

* absence of PH
* absence of RV diastolic dysfunction by echo
* RV systolic dysfunction
* age < 18 years
* contraindication to MRI
* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: specialist clinics community
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Correlation between RV diastolic function and vorticity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Brett Fenster, MD, FACC, FACP, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Background] Shiina Y, Funabashi N, Lee K, Daimon M, Sekine T, Kawakubo M, Sekine Y, Takahashi M, Yajima R, Wakatsuki Y, Tanabe N, Kuriyama T, Komuro I. Doppler imaging predicts cardiac events in chronic pulmonary thromboembolism. Int J Cardiol. 2009 Apr 3;133(2):167-72. doi: 10.1016/j.ijcard.2007.12.017. Epub 2008 Feb 1. PMID 18242738
- [Background] Shiina Y, Funabashi N, Lee K, Daimon M, Sekine T, Kawakubo M, Takahashi M, Yajima R, Tanabe N, Kuriyama T, Komuro I. Right atrium contractility and right ventricular diastolic function assessed by pulsed tissue Doppler imaging can predict brain natriuretic peptide in adults with acquired pulmonary hypertension. Int J Cardiol. 2009 Jun 12;135(1):53-9. doi: 10.1016/j.ijcard.2008.03.090. Epub 2008 Sep 14. PMID 18793807
- [Background] Pasipoularides AD, Shu M, Womack MS, Shah A, Von Ramm O, Glower DD. RV functional imaging: 3-D echo-derived dynamic geometry and flow field simulations. Am J Physiol Heart Circ Physiol. 2003 Jan;284(1):H56-65. doi: 10.1152/ajpheart.00577.2002. Epub 2002 Sep 12. PMID 12388220
- [Background] Kheradvar A, Gharib M. On mitral valve dynamics and its connection to early diastolic flow. Ann Biomed Eng. 2009 Jan;37(1):1-13. doi: 10.1007/s10439-008-9588-7. Epub 2008 Nov 4. PMID 18982451
- [Background] Hong GR, Pedrizzetti G, Tonti G, Li P, Wei Z, Kim JK, Baweja A, Liu S, Chung N, Houle H, Narula J, Vannan MA. Characterization and quantification of vortex flow in the human left ventricle by contrast echocardiography using vector particle image velocimetry. JACC Cardiovasc Imaging. 2008 Nov;1(6):705-17. doi: 10.1016/j.jcmg.2008.06.008. Epub 2008 Nov 18. PMID 19356506